CLINICAL TRIAL: NCT06066333
Title: Safety and Immunological Effects of Pembrolizumab Plus Ablative Radiotherapy in Patients With Advanced Adrenocortical Carcinoma
Brief Title: Study of Radiotherapy and Pembrolizumab in People With Adrenocortical Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-272
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Adrenocortical Carcinoma; ACC; Metastatic Adrenocortical Carcinoma
Keywords: Adrenocortical Carcinoma; ACC; Metastatic Adrenocortical Carcinoma; Metastatic ACC; Metastatic ACC with symptomatic liver metastases; 23-272; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Adrenocortical Carcinoma (Experimental): Participants with histologically proven metastatic Adrenocortical Carcinoma/ACC with both intra-hepatic and extra-hepatic sites of disease.
  Interventions: Radiation: Ablative Radiotherapy; Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Ablative Radiotherapy — All participants will first undergo ablative RT
  Other Names: Ablative RT
Drug: Pembrolizumab — After completion of ablative RT, all subjects may begin pembrolizumab treatment

SUMMARY:
The purpose of this study is to determine whether pembrolizumab given after standard ablative Radiotherapy is a safe treatment that causes few or mild side effects in people with advanced Adrenocortical Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be ≥ 15 years of age on day of signing informed consent.
* Have histologically- or cytologically- confirmed metastatic ACC with symptomatic liver metastases.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or
* Adequate performance status:

  1. Patients < 16 years of age: Lansky ≥ 50%
  2. Patients ≥ 16 years of age: Karnofsky ≥ 50%
* Have measurable disease based on RECIST v1.1.
* Have radiologic documentation of extrahepatic tumor, defined as extrahepatic metastases.
* Consent for use of archived tissue for research purposes. Archival tissue (1 block or 20 unstained slides) will be requested, when available.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 28 days of treatment initiation.

Table 1: Adequate Organ Function Laboratory Value

Hematological Absolute neutrophil count (ANC) ≥1,500 / mcL Platelets ≥100,000 / mcL

Renal Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

*Creatinine clearance should be calculated per institutional standard.

Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 5 X ULN

Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

* Female subjects of childbearing potential should have a negative serum pregnancy test within 72 hours prior to beginning treatment on study. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 10.6.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free of menses for >1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to study Day 1 (the first day of ablative RT).
* Has undergone radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields (to include Y90).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study Day 1. The use of physiologic doses of corticosteroids for adrenal and pituitary insufficiency is not considered a form of systemic steroid therapy and would not exclude a subject from the study.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. The use of non-immunotherapy monoclonal antibodies (such as dupilumab (for eczema), omalizumab (for urticaria), benralizumab (for asthma)) would not exclude a subject from the study.
* Has had prior chemotherapy, targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

Note: Subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.

* If subject underwent major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to beginning treatment on study and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for brain metastases for at least 7 days prior to study Day 1. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study. Subjects that have adrenal or pituitary insufficiency that require physiologic corticosteroid replacement therapy would not be excluded from the study. Subjects who are on mitotane for control of hormonal symptoms for their disease at the time of eligibility assessment can continue on mitotane during the course of the study.
* Has evidence of interstitial lung disease or history of (non-infectious) pneumonitis that required steroids or current pneumonitis. 11. Has an active infection requiring systemic therapy. 12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. 13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial. 14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to study Day 1. Administration of killed vaccine is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-09-27 (Estimated); Study Completion 2026-09-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants evaluated for AEs | up to 1 year
  The primary objective of this pilot study is to evaluate the safety of treatment with ablative Radiotherapy/RT followed by pembrolizumab in patients with advanced Adrenocortical Carcinoma/ACC by evaluating treatment related adverse events. AEs will be recorded according to "Common Terminology Criteria for Adverse Events" v5.0 (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Nitya Raj, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack, Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org